CLINICAL TRIAL: NCT03884933
Title: Large Scale Implementation of Community Based Mental Health Care for People With Severe and Enduring Mental Ill Health in Europe
Acronym: RECOVER-E
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Enrolling by invitation
Sponsor: Liga Romana pentru Sanatate Mintala (Other)
Collaborators: Psychiatric Hospital for Chronic Patients Siret, Suceava, Romania (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Supportive Care
Other Study IDs: 779362
Record Dates: First submitted 2019-03-20; First posted 2019-03-21 (Actual); Last update posted 2019-05-16 (Actual); Status verified 2019-03

CONDITIONS: Mental Disorders, Severe
MeSH Terms: conditions — Mental Disorders

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Mobile team community mental health services (Experimental)
  Interventions: Other: Mobile team community mental health services
- Current clinical services (No Intervention)

INTERVENTIONS:
Other: Mobile team community mental health services — The intervention focuses on changing mental health care systems to be able to provide community-based mental health care for people with severe mental illness. This will be done through the development and implementation of multidisciplinary community mental health teams (CMHTs) in each of the implementation sites, consisting of at least one nurse, psychiatrist, psychologist, social worker, and peer worker (person with lived experience of a severe mental illness). The structure and delivery method of the community mental health teams is part of an evidence-based service delivery model providing flexible, assertive community mental health teams providing integrated services to people with severe mental illness (SMI) in order to structurally attain their recovery goals, as well as timely and appropriate care in the event of a crisis.
  Arms: Mobile team community mental health services

SUMMARY:
RECOVER-E's main purpose is to ensure well-functioning community mental health teams in five countries in Europe; these teams will serve as the central node for the coordination and provision of care for people with severe mental illness (SMI). At present, specialist teams providing comprehensive, evidence-based mental health care are not available or functional in many countries in Eastern Europe, and the care pathways and evidence-based treatment protocols for community-based and recovery-oriented mental healthcare have not been defined or tailored to local situations and therefore, are not being implemented. This project aims to implement and study community-based initiatives to narrow this gap. These efforts will emphasize the development of human resource capacity and care pathways that can be distilled in a comprehensive pathway to scale for regional and national decision-makers for potential project expansion and replication after the project period.

DETAILED DESCRIPTION:
AIMS / OBJECTIVES The overall aim of Recover-E is to contribute to the implementation of a community-based service delivery model in five implementation sites in low and middle-income countries and vulnerable populations in high-income countries in Europe to improve the level of functioning, quality of life, and mental health outcomes for people with severe and enduring mental ill health (schizophrenia, bipolar disorder, depression).

RECOVER-E's specific project objectives are to:

* design, implement and evaluate recovery-oriented care for people with severe mental illness in community settings by recognizing the value of experiential knowledge through including peer experts as members of the community mental health teams
* identify intervention and program elements, as well as contextual factors, which enhance sustainable implementation of community-based mental healthcare for people with severe mental illness
* establish a peer-to-peer capacity building partnership in community mental health, by linking a European expert panel with key stakeholders in five implementation sites (policy makers, service managers, service providers, users, and carers) to co-create community health services for people with SMI
* develop evidence-based care pathways and treatment protocols and transition to scale for regional and national decision-makers, for continued implementation and scale up after the project's life span

ELIGIBILITY:
Inclusion Criteria:The target population for inclusion in the study are consenting adults (ages 18-65 years) with severe mental illness (SMI), defined based on Deslespaul's conceptualisation of SMI:

1. meets criteria for (and presence of) bipolar disorder, severe major depression, schizophrenia, schizophreniform, and schizoaffective disorder according to the International Statistical Classification of Diseases and Related Health Problems (ICD-10). The person should require care and treatment and not be in symptomatic remission;
2. has severe limitations in social and community functioning;
3. problems are not transient in nature; the problems are systematic and long-term, and potentially chronic, intermitted, and/or recurrent;
4. coordinated care provided by care networks or multidisciplinary teams is needed to deliver treatment
5. Patients with prevalence of suicidal behaviours (including suicide attempts)

Exclusion criteria are:

1. Patients under the age of 18
2. Patients with dementia or Alzheimer's disease
3. Patients for whom treatment is legally prescribed (in forensic psychiatry), however if they are discharged from the forensic ward, and still in need of treatment they can be included

Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 180 (Estimated)
Dates: Start 2019-03-01 (Actual); Primary Completion 2020-12-01 (Estimated); Study Completion 2020-12-31 (Estimated)

PRIMARY OUTCOMES:
The primary outcome is global (personal and social) functioning, measured with the World Health Organization Disability Assessment Schedule 2.0 (WHODAS 2.0). | 18 months
  The WHODAS 2.0 is a generic measure designed to measure functioning and disability as well as health-related quality of life based on the Internal Classification of Functioning (ICF) framework. The WHODAS 2.0 will be used as a continuous outcome in the clinical trial evaluation. The scale comes in 12- and 36-item versions. The 36-item version captures the level of functioning in six domains of life:
  Domain 1: Cognition - understanding and communicating Domain 2: Mobility - moving and getting around Domain 3: Self-care - attending to one's hygiene, dressing, eating and staying alone Domain 4: Getting along - interacting with other people Domain 5: Life activities - domestic responsibilities, leisure, work and school Domain 6: Participation - joining in community activities, participating in society
  The 12-item version helps to assess overall (global) functioning only. Therefore, it is planned to use the 36-itme self-report version of the WHODAS 2.0.

CONTACTS AND LOCATIONS:
Locations (1):
- Spitalul de Psihiatrie Cronici Siret, Siret, Suceava, Romania

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Shields-Zeeman L, Smit F, Wijnen B, Roth C, Wensing M, Petrea I; RECOVER-E consortium; Bolinski F, Bajraktarov S, Dedovic J, Keet R, Rojnic Kuzman M, Nakov V, Nica R, Novotni A, Tomcuk A, Djurisic T, Morales G, Rotaru Anghelescu T; RECOVER-E study. Community versus institutionalised care for people with severe mental illness in five countries in Southeast Europe: pooled analysis of five randomised trials. BMJ Glob Health. 2025 Oct 23;10(10):e018594. doi: 10.1136/bmjgh-2024-018594. PMID 41130742
- [Derived] Roth C, Wensing M, Kuzman MR, Bjedov S, Medved S, Istvanovic A, Grbic DS, Simetin IP, Tomcuk A, Dedovic J, Djurisic T, Nica RI, Rotaru T, Novotni A, Bajraktarov S, Milutinovic M, Nakov V, Zarkov Z, Dinolova R, Walters BH, Shields-Zeeman L, Petrea I. Experiences of healthcare staff providing community-based mental healthcare as a multidisciplinary community mental health team in Central and Eastern Europe findings from the RECOVER-E project: an observational intervention study. BMC Psychiatry. 2021 Oct 24;21(1):525. doi: 10.1186/s12888-021-03542-2. PMID 34689733
- [Derived] Wijnen BFM, Smit F, Uhernik AI, Istvanovic A, Dedovic J, Dinolova R, Nica R, Velickovski R, Wensing M, Petrea I, Shields-Zeeman L. Sustainability of Community-Based Specialized Mental Health Services in Five European Countries: Protocol for Five Randomized Controlled Trial-Based Health-Economic Evaluations Embedded in the RECOVER-E Program. JMIR Res Protoc. 2020 Jun 1;9(6):e17454. doi: 10.2196/17454. PMID 32476658